CLINICAL TRIAL: NCT00600574
Title: A Randomized Controlled Trial Comparing the Efficay and Tolerability of Ai Chi Versus Stretching in Fibromyalgia Management: a Six Months Study
Brief Title: Ai Chi Versus Stretching in Fibromyalgia Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Elena Pita Calandre, Professor of Pharmacology, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML-2007
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; physical therapies; stretching; Ai Chi
MeSH Terms: conditions — Fibromyalgia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S (Active Comparator): physiotherapy in warm pool by means of stretching
  Interventions: Other: physical therapy
- AI (Experimental): physiotherapy in warm pool by means of Ai Chi
  Interventions: Other: physical therapy

INTERVENTIONS:
Other: physical therapy — weekly pool physiotherapy with muscle stretching
  Other Names: physiotherapy
  Arms: S
Other: physical therapy — weekly pool physiotherapy with Ai Chi movements during a 6 months period
  Other Names: physiotherapy
  Arms: AI

SUMMARY:
The purpose of the study is to compare the efficacy and tolerability of Ai Chi, an adaptation of Tai Chi exercise to water, with stretching on fibromyalgia symtomatology.

DETAILED DESCRIPTION:
Physical therapies have shown to be effective in the treatment of fibromyalgia and It is generally assumed that a multidisciplinary approach, combining both pharmacologic and non-pharmacologic measures, is probably the optimal treatment approach for most fibromyalgia patients. As these patients are usually physically deconditioned, low-intensity exercise has been recommended at least as initial treatment. At this respect, exercise in warm water is considered a good option as both temperature and water buoyancy minimize body weight's stress and help patients to minimize pain. In a previous study comparing short term physiotherapy with stretching and Ai Chi we found that Ai Chi was at least as effective as stretching and induced a significant reduction in fibromyalgia core symptomatology and in sleep parameters. The objective of the present randomized controlled study is to compare both physiotherapy techniques in a long term basis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of fibromyalgia according to the ACR criteria
* 18 years or older
* written informed consent to participate

Exclusion Criteria:

* unable to tolerate warm chlorinated water
* associated medical condition contraindicating exercise in warm water

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Fibromialgya Impact Questionnaire | baseline, 6 months, 1 year

SECONDARY OUTCOMES:
Pittsbugh Sleep Quality Index | baseline, 6 months, 12 months
Hospital Anxiety and Depression Scale | baseline, 6 months, 12 months
SF-36 Health Survey | baseline, 6 months, 12 months
Brief Pain Inventory | baseline, 6 months, 12 months
Adverse reaction recording | baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elena P. Calandre, M.D., Study Director — Universidad de Granada
Locations (1):
- Hospital Universitario "Virgen de las Nieves", Granada, Granada, Spain

REFERENCES:
- [Background] Gowans SE, deHueck A. Pool exercise for individuals with fibromyalgia. Curr Opin Rheumatol. 2007 Mar;19(2):168-73. doi: 10.1097/BOR.0b013e3280327944. PMID 17278933